CLINICAL TRIAL: NCT04852159
Title: Test of Reliability and Validity of the Cerebral Palsy Quality of Life Questionnaire in Local Languages of Pakistan.
Brief Title: Translation of the Cerebral Palsy Quality of Life Questionnaire in Local Languages of Pakistan.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00959 Gul Andama
Record Dates: First submitted 2021-04-10; First posted 2021-04-21 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy
Keywords: CP, cerebral palsy, children, quality of life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive analytical study to translate the CP-QOL into local languages of Pakistan that are, Pashto, Urdu, Punjabi, Sindhi and Balochi languages. Along with validation of the translated versions by evaluating their validity and reliability in the people of Pakistan, speaking respective languages and suffering from low back pain. No such study has been previously conducted in the Pakistan region which translates the scale and follows the proper cross-culture adaptation.

Condition or disease: Cerebral palsy. Non-probability Purposive Sampling would be used. The study will be conducted in relevant areas of Pakistan.

DETAILED DESCRIPTION:
CP QOL has two separate forms, for both the child and the primary caregiver. CP QOL- The primary caregiver proxy report consists of 66 items for children ages 4-12 years old.

The child self-report form contains 52 items for children ages 9-12 years old. The version CP QOL-Child Self Report Questionnaire (9-12 years) is divided into areas: well-being and social acceptance, functionality, participation and physical health, emotional well-being and self-esteem, access to services and pain and impact disability.

This version should be answered by the children with CP, that is, it is the child's self-report.

All the items are rated from 1 to 9, except for one item in pain and impact of disability domain, which is rated on a 5-point scale. All responses will then be converted into scale score between 0 to 100. Higher scores meant a higher quality of life. In case children needed any help while filling out the questionnaires, they could easily consult caregivers or researchers. As the CP QOL-Child is a well-developed measurement scale, it is meaningful to validate its Urdu, Pushto, Punjabi, Sindhi and Balochi versions. It is also useful to study the QOL of children with CP in different cultural settings by using the same measurement items so that a more direct comparison can be made. Therefore, the aim of this study is to translate the CP QOL questionnaire in Urdu, Pushto, Punjabi, Sindhi and Balochi and also to assess the reliability and validity of this translated version of CP QOL questionnaire in Pakistan.

The translation and cultural adaptation processes would start after obtaining approval from the developer of the original CP QOL Child. This would be done according to WHO guidelines. Translation will be done by symmetrical category. The purpose will be to gain uniformity in the translation of tool in both the Target language and Source language. This will involve 5 steps. (Forward translation, synthesis 1, Back translation, synthesis 2 and pilot testing.) Phase 2 would be done according to the guidelines of COSMIN in which psychometric properties will be measured. (reliability, internal consistency, construct validity and factor analysis.)

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9 to 12 years.

  * Children who are diagnosed with cerebral palsy.
  * Children who are able to read.

Exclusion Criteria:

* Children suffering from neurodegenerative diseases or psychiatric illness

Ages: 9 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: 525
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-04-22 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
CP QOL Child Self report version. | 8 months
  The child self-report form contains 52 items for children ages 9-12 years old. The version CP QOL-Child Self Report Questionnaire (9-12 years) is divided into areas: well-being and social acceptance, functionality, participation and physical health, emotional well-being and self-esteem, access to services and pain and impact disability.
  All the items are rated from 1 to 9, except for one item in pain and impact of disability domain, which is rated on a 5-point scale. All responses will then be converted into scale score between 0 to 100. Higher scores meant a higher quality of life. In case children needed any help while filling out the questionnaires, they could easily consult caregivers or researchers. The total score is 100, the minimum score is 0 and the maximum score is 100.

SECONDARY OUTCOMES:
Reliability of translated versions of CP QOL Child | 8 months
  To determine the reliability of cross-culturally adapted and translated CP-QOL Child in children having cerebral palsy of respective languages. Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two intervals between different visits of the patient. Thus this will be measured through test re-test reliability.
Validity of translated versions of CP QOL Child | 8 months
  To determine the validity of cross-culturally adapted and translated CP-QOL Child in children having cerebral palsy of respective languages. Validity is how accurate the results are. Thus this will be measured through various parameters to validate the translated versions as appropriate and applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Ali Muhammad Memorial, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Development and exploration of a Japanese version of the cerebral palsy quality of life for children questionnaire for primary caregivers: a pilot study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6751053/
- See also: Quality of life of Finnish children with cerebral palsy — https://pubmed.ncbi.nlm.nih.gov/26119576/
- See also: A quality of life questionnaire for adolescents with cerebral palsy: psychometric properties of the Bengali CPQoL-teens — https://hqlo.biomedcentral.com/articles/10.1186/s12955-019-1206-x